CLINICAL TRIAL: NCT02778152
Title: Pilonidal Disease Laser Depilation Pilot Study
Brief Title: Pilot Study of Laser Hair Depilation for Pilonidal Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Minneci (Other)
Responsible Party: Sponsor-Investigator, Peter Minneci, Principal Investigator, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-00104
Record Dates: First submitted 2016-05-17; First posted 2016-05-19 (Estimated); Results first posted 2019-03-26 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-03

CONDITIONS: Pilonidal Disease

STUDY DESIGN:
Intervention Model Description: Laser hair removal
Oversight: Data Monitoring Committee: No

ARMS (1):
- Laser depilation (Experimental): Laser depilation to the natal cleft (pilonidal region) monthly for 5 treatments with either an 810nm of Nd:YAG laser dependent on Fitzpatrick skin type and tolerability.
  Interventions: Device: Laser depilation

INTERVENTIONS:
Device: Laser depilation — Laser depilation of natal cleft (pilonidal region)

SUMMARY:
Pilot study to assess tolerability and safety of laser hair depilation in adolescents and young adults with pilonidal disease.

DETAILED DESCRIPTION:
This is a pilot study to measure safety and tolerance of laser hair depilation in adolescents and young adults with pilonidal disease as a potential treatment to intervene on future recurrence.

Up to a total of 10 patients will be enrolled.

Each patient will be involved in the study for one year. Patients will be brought into Surgery clinic for 1 laser treatment every 4-6 weeks to obtain a total of 5 treatments. Follow up will occur monthly from the time of initial treatment through 1 year after the last treatment as we evaluate for tolerance and efficacy.

Inclusion Criteria

* English and non-English speaking patients
* All Fitzpatrick skin types
* Age : 12-20 years
* Diagnosis of pilonidal disease

Exclusion Criteria

* History of photosensitivity
* Actively inflamed pilonidal sinus

Laser depilation treatment: Patients will be brought into Surgery clinic for 1 treatment every 4-6 weeks to obtain a total of 5 treatments. The treatment will consist of an 810 nm or Nd:YAG depending on Fitzpatrick skin type and tolerability. A cooling platform and application of topical lidocaine cream will be used to minimize any discomfort associated with the heat of the laser treatments.

Initial follow up for the laser depilation group will be performed to assess for tolerance of the laser treatment. Patients will report their pain every 6 hours for the first 48 hours after their laser hair depilation treatment. Once tolerance is established, patients will return to surgical clinic every month for their laser or placebo visit. After the 5th clinic visit, they will receive a telephone call monthly to assess for any evidence of resolution or recurrence of disease up to 1 year after the completion of the treatments.

ELIGIBILITY:
Inclusion Criteria:

* English and non-English speaking patients
* All Fitzpatrick skin types
* Age : 12-20 years
* Diagnosis of pilonidal disease

Exclusion Criteria:

* History of photosensitivity
* Actively inflamed pilonidal sinus

Ages: 12 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2016-02-19 (Actual); Primary Completion 2018-02-02 (Actual); Study Completion 2018-02-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter C Minneci, MD, Principal Investigator — Research Institute at Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Laser Group: Received 5 laser hair removal treatments spaced every 4 to 6 weeks
Period: Overall Study
Arm/Group | Laser Group
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Not applicable--- units analyzed are participants
Arm/Group | Laser Depilation
Number analyzed (Participants) | 13
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 16.6 [14 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 11
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of Laser Treatment
Description: Median of pain scores immediately post-laser treatment after each of the 5 treatments. Pain was assessed on a scale of 1 to 10, 10 being the greatest amount of pain.
Time Frame: five months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Laser Group
Number analyzed (Participants) | 13
score on a scale | 2 [2 to 2]

2. Secondary Outcome: Number of Participants Experiencing Second Degree Burns Post-Treatment
Description: Incidence of skin burn within the first 48 hours after each of the 5 treatments
Time Frame: five months
Measure: Count of Participants; unit: Participants
Arm/Group | Laser Group
Number analyzed (Participants) | 13
Participants | 0

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Laser Group
All-Cause Mortality (participants affected / at risk) | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13
Other Adverse Events (participants affected / at risk) | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT02778152/Prot_SAP_000.pdf